CLINICAL TRIAL: NCT05072691
Title: Prognostic Value of Cerebrospinal Fluid Immunoglobulin Free Light Chains in Patients With Multiple Sclerosis
Status: Recruiting | Type: Observational
Sponsor: Francis Corazza (Other)
Responsible Party: Sponsor-Investigator, Francis Corazza, Head of Immunology laboratory, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Other Study IDs: CHUB-Neuro-Lab-MS
Record Dates: First submitted 2021-09-13; First posted 2021-10-11 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood and cerebrospinal fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Patients with Multiple sclerosis and Optic Neuritis: Patients ≥ 18 year-old at the time of enrollment, with newly diagnosed multiple sclerosis according to 2017 McDonald diagnostic criteria Patients ≥ 18 year-old at the time of enrollment with first episode of optic neuritis, fulfilling or not (i.e. CIS, clinically isolated syndrome) 2017 McDonald diagnostic criteria for multiple sclerosis
  Interventions: Diagnostic Test: CSF immunoglobulin (Ig) free light chains (FLC) dosage
- Patients with non-inflammatory neurologic diseases (NIND): Patients ≥ 18 year-old with suspected non-inflammatory neurologic diseases (such as Alzheimer disease, intracranial hypertension, etc) receiving routine diagnostic lumbar puncture
  Interventions: Diagnostic Test: CSF immunoglobulin (Ig) free light chains (FLC) dosage
- Patients with other inflammatory neurologic diseases (IND): Patients ≥ 18 year-old with suspected inflammatory neurologic diseases other than multiple sclerosis (such as inflammatory peripheral neuropathies, meningitis, neuromyelitis optica spectrum disorders, etc) receiving routine diagnostic lumbar puncture
  Interventions: Diagnostic Test: CSF immunoglobulin (Ig) free light chains (FLC) dosage

INTERVENTIONS:
Diagnostic Test: CSF immunoglobulin (Ig) free light chains (FLC) dosage — CSF immunoglobulin (Ig) free light chains (FLC) dosage in the peripheral blood and cerebrospinal fluid.

SUMMARY:
Multiple sclerosis (MS) is a chronic inflammatory autoimmune disease of the central nervous system, usually presenting as clinically isolated syndrome (CIS). The course of MS following first symptoms is unpredictable, as approximately 30% of patients with MS have a benign course and don't develop significant disability while another 20-30% progress to severe disability within a relatively short time period. In this context, it is difficult to counsel an individual patient and choose the best treatment option at time of diagnosis. For these reasons, prognostic markers that could be used to predict future disease course are extremely useful.

The only cerebrospinal fluid (CSF) prognostic biomarker currently used in clinical practice are oligoclonal bands (OCB) that can predict conversion from CIS to clinically definite MS, although this observation is not consistent. However, OCB analyses are qualitative with issues in reproducibility and a limited dynamic range. CSF immunoglobulin (Ig) free light chains (FLC) are a quantitative measure of humoral response in CSF that has showed greater sensitivity and specificity than OCB for confirming diagnosis of MS. Moreover, in few recent studies they seem to have also a prognostic value, predicting conversion from CIS to clinically definite MS and correlating with the Expanded Disability Status Scale (EDSS).

Optic Neuritis (ON) can be a first clinical relapse of MS and is particularly interesting because it may constitute a suitable clinical model for neuroprotection studies, as visual function can be measured with quantitative methods, including Visual Evoked Potential (VEP) and Optical Coherence Tomography (OCT).

The investigators aim to better explore the utility of CSF Ig FLC as potential prognostic biomarker for MS, and to predict the recovery of visual function after ON, as model of MS relapse.

The investigators will study its potential correlation with MS relapses, with changes in several functional outcome scores, exploring physical disability, fatigue, behavior, cognition, upper and lower extremity function, and with MRI disease activity. For a subgroup of patient, the investigators aim to explore its potential correlation with in vivo measures of demyelination and neuronal and axonal loss after ON, as model of potential recovery after MS relapse. The investigators aim also to compare the prognostic value of Ig FLC with Neurofilament light chain (NfL), a potential prognostic biomarker wider studied in MS.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic inflammatory autoimmune disease of the central nervous system, usually presenting as clinically isolated syndrome (CIS). The course of MS following first symptoms is unpredictable, as approximately 30% of patients with MS have a benign course and don't develop significant disability while another 20-30% progress to severe disability within a relatively short time period. In this context, it is difficult to counsel an individual patient and choose the best treatment option at the time of diagnosis. For these reasons, prognostic markers that could be used to predict future disease course are extremely useful.

The only cerebrospinal fluid (CSF) prognostic biomarker currently used in clinical practice are oligoclonal bands (OCB), that can predict the conversion from CIS to clinically definite MS, although this observation is not consistent. However, OCB analyses are qualitative, with issues in reproducibility and a limited dynamic range.

CSF immunoglobulin (Ig) free light chains (FLC) are a quantitative measure of humoral response in CSF that had shown greater sensitivity and specificity than OCB for confirming diagnosis of MS. Moreover, in few recent studies, they showed to have also a potential prognostic value, predicting conversion from CIS to clinically definite MS and correlating with the Expanded Disability Status Scale (EDSS), a scale widely used in clinical practice as marker of MS disability. However, this scale counts very close to ambulation abilities and poorly correlates with other frequent MS symptoms, such as upper extremity disability, fatigue, cognitive and neuropsychiatric symptoms.

One of the most currently studied biomarkers of disease activity and treatment response in MS, not yet widely available in clinical practice, is represented by Neurofilament light chain (NfL). Elevated CSF and blood concentrations of NfL were found to correlate with an increase in the number of relapses, disability worsening, MRI disease activity, and brain volume loss in MS. Blood NfL was shown to strongly correlate with NfL in the CSF of patients with MS and has been proposed as an easily accessible biomarker of treatment response.

Optic Neuritis (ON) can be a first clinical manifestation of MS and is particularly interesting since it may constitute a suitable clinical model for neuroprotection studies. First, visual function can be measured with quantitative methods, including low-contrast acuity, visual fields, and color discrimination. Secondly, Visual Evoked Potential (VEP) with the evaluation of P100 latency, and Optical Coherence Tomography (OCT) with the evaluation of Ganglion Cell Layer (GCL) and Retinal Nerve Fiber Layer (RNFL) thickness, represent in-vivo measures of demyelination, and neuronal and axonal loss secondary to ON, respectively. The investigators aim to better explore the utility of CSF Ig FLC as potential prognostic biomarker of disease activity, disability worsening, and treatment response in patients with MS, and as potential predictor of visual recovery after ON as model of MS relapse. To investigate the prognostic value of CSF Ig FLC, the investigators evaluate the correlation of CSF Ig FLC at the time of MS diagnosis with clinical relapse, with changes in several functional outcome scores, exploring physical disability, fatigue, behavior, cognition, upper and lower extremity functions, and with MRI disease activity. For a subgroup of patient, the investigators aim to explore the correlation of CSF Ig FLC with in vivo measures of demyelination, neuronal and axonal loss after ON, as model of potential recovery after MS relapse. The investigators aim also to compare the prognostic value of Ig FLC with Neurofilament light chain (NfL) concentrations in CSF and blood.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 at the time of enrollment
* Diagnosis of multiple sclerosis according to 2017 McDonald diagnostic criteria or optic neuritis (fulfilling or not criteria for multiple sclerosis, i.e. clinically isolated syndrome)
* Receiving both lumbar puncture and brain MRI for the routine diagnostic work-up

Exclusion Criteria:

• None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients with MS and ON
  * Patients with non-inflammatory neurologic diseases (NIND) and patients with other inflammatory neurologic diseases (IND) as control group
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-07-14 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Expanded Disability Status Scale (EDSS) | Change from baseline (time of enrollment) up to 4 years
  Ordinal scale of 0.0-10 ("no disability" to "death due to MS"), with higher scores reflecting greater level of disability.
Fatigue Severity Scale (FSS) | Change from baseline (time of enrollment) up to 4 years
  Frequently used nine-item questionnaire for the evaluation of fatigue in patients with MS (10). The FSS score is the mean score of the nine items with a cut-off for fatigue set to ≥ 4.
Hospital Anxiety and Depression Scale (HADS) | Change from baseline (time of enrollment) up to 4 years
  The scale is a 14-item self-report measure with seven items each in the depression and anxiety subscales. Each item was scored on a scale of 0-3, with a total potential score of 21, where a threshold score of 8 or greater on each subscale is considered indicative of clinically significant anxiety or depression.
Symbol-Digit Modalities Test (SDMT) | Change from baseline (time of enrollment) up to 4 years
  The test consists of a series of single digits paired with nine symbols, as a reference key. The patient views a pseudorandomized sequence of these symbols and orally responds with the matching digit. The final score is the number of correct responses within 90 seconds, with higher scores corresponding to faster processing speed.
Nine Hole Peg Test (NHPT) | Change from baseline (time of enrollment) up to 4 years
  Brief, standardized, quantitative test, where the patient picks up nine pegs one at a time as quickly as possible, puts them in nine holes, and, once they are in the holes, removes them again as quickly as possible one at a time, replacing them into a container. The total time to complete the task is recorded. Two consecutive trials with the dominant hand are immediately followed by two consecutive trials with the non-dominant hand. The final score is an average of the four trials.
Timed 25-Foot Walk (T25FW) | Change from baseline (time of enrollment) up to 4 years
  Quantitative mobility and leg function performance test where the patient is instructed to walk 25 feet as quickly as possible. The time is calculated from the initiation of the instruction to start and ends when the patient has reached the 25-foot mark. The task is immediately administered again by having the patient walk back the same distance. The score is the average of time for the two completed trials.
Six Spot Step Test (SSST) | Change from baseline (time of enrollment) up to 4 years
  The patient is instructed to walk as quickly as possible from one end to the other of a rectangular field measuring 1 x 5 m, while kicking five cylinder blocks out of five circles marked on the floor. The patient has to do four runs, two for each leg. The total score of the SSST is the mean value of time used for each of the four runs.
Ambulation Score (AS) | Change from baseline (time of enrollment) up to 4 years
  The AS is the measure of the distance the patient is able to walk in meters. The score ranges from 0 (ambulation unrestricted) to 12 (essentially restricted to bed).
Annualized relapse rate (ARR) | Once a year during the observational period.
  Number of relapses per year from disease onset
MRI data: T2 lesions | Change from baseline (time of enrollment) up to 4 years
  T2 lesion load in brain and spinal cord
MRI data : gadolinium enhancing lesions | Change from baseline (time of enrollment) up to 4 years
  Gadolinium enhancing lesions in brain and spinal cord
P100 latency (VEP) | Change from baseline (time of enrollment) up to 4 years
  VEP is a measurement of the electrical signal recorded at the scalp over the occipital cortex in response to light stimulus. The studied VEP contains an initial negative peak (N1), followed by a positive peak (P100). Demyelination of the optic nerve results in increased latency of the P100 waveform, without significant effect on amplitude.
Visual acuity | Change from baseline (time of enrollment) up to 4 years
  Low-contrast letter acuity chart measured by low-contrast Sloan letter chart.
Visual field | Change from baseline (time of enrollment) up to 4 years
  Visual field measured by 30-2 SITA Standard visual field test
Color discrimination | Change from baseline (time of enrollment) up to 4 years
  Color discrimination measured by Ishihara test
GCL thickness (OCT) | Change from baseline (time of enrollment) up to 4 years
  OCT is a technique using light waves to take cross-section pictures of retina. It allows measuring of thickness of different retinal layer. The anterior visual pathways consist of the retinal ganglion cells, whose somas are in the ganglion cell layer (GCL) and axons form the retinal nerve fiber layer (RNFL). Assessment of the RNFL and GCL using OCT potentially allows assessing of axonal and neuronal degeneration.
RNFL thickness (OCT) | Change from baseline (time of enrollment) up to 4 years
  OCT is a technique using light waves to take cross-section pictures of retina. It allows measuring of thickness of different retinal layer. The anterior visual pathways consist of the retinal ganglion cells, whose somas are in the ganglion cell layer (GCL) and axons form the retinal nerve fiber layer (RNFL). Assessment of the RNFL and GCL using OCT potentially allows assessing of axonal and neuronal degeneration.
immunoglobulin (Ig) free light chains (FLC) | Baseline
  Ig FLC concentrations will be measured using the Freelite Mx (CSF) assay (The Binding Site Group, Bimingham, UK) in the peripheral blood and cerebrospinal fluid.

CONTACTS AND LOCATIONS:
Overall Officials: Serena Borrelli, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No